CLINICAL TRIAL: NCT03442530
Title: Tobacco Use in Pregnancy Intervention for Cessation
Acronym: ToPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristin Ashford (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Kristin Ashford, Associate Dean of Undergraduate Faculty Affairs, University of Kentucky College of Nursing, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0658-P3K
Record Dates: First submitted 2018-01-30; First posted 2018-02-22 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy
Keywords: pregnancy, smoking cessation, tobacco, preterm birth, ToPIC
MeSH Terms: conditions — Smoking Cessation; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobacco Treatment As Usual (TTAU) (Active Comparator): Eligible women assigned to the control group will be informed of the risks of tobacco use and benefits of quitting using the ACOG 5A's approach by their healthcare provider.5 This standard takes approximately 5-15 minutes, and is offered at each prenatal and postpartum appointment. The study coordinator will invite participants to complete the tobacco use questionnaires (TUQ),urine cotinine validation, and Expired Air Carbon Monoxide (EACO) analysis to assess ongoing tobacco use at the designated time points.
  Interventions: Behavioral: Tobacco Treatment As Usual (TTAU)
- ToPIC (Experimental): Eligible women assigned to the intervention will receive TTAU plus ToPIC administered by the CTTS. At least once monthly, at routinely scheduled prenatal visits or through telephone, the CTTS will provide cessation counseling. The CTTS will invite participants to complete TUQs,urine cotinine validation and EACO analysis to assess ongoing tobacco use at the designated time points.
  Interventions: Behavioral: ToPIC

INTERVENTIONS:
Behavioral: ToPIC — Expanded tobacco cessation counseling for pregnant women.
  Arms: ToPIC
Behavioral: Tobacco Treatment As Usual (TTAU) — Standard of care tobacco cessation counseling for pregnant women
  Arms: Tobacco Treatment As Usual (TTAU)

SUMMARY:
The proposed project will test the effectiveness of the novel delivery of an established tobacco cessation treatment among pregnant women in Kentucky. Tobacco use during pregnancy is one of the most modifiable risk factors associated with poor birth and maternal outcomes and yet smoking prevalence among pregnant women in Kentucky is among the highest in the county and estimated to be twice that of the national average, with no meaningful declines observed in twenty years.

DETAILED DESCRIPTION:
The purpose of this pilot project is to test effectiveness of a tobacco-treatment cessation intervention (American College of Obstetricians and Gynecologists (ACOG) 5 A's) through use of a non-physician healthcare champion from within the clinic's existing infrastructure. This Tobacco use in Pregnancy Intervention for Cessation (ToPIC) will involve training the identified healthcare provider to become a Certified Tobacco Treatment Specialist (CTTS) and to administer the 5 A's to pregnant Medicaid patients receiving prenatal care through two high-volume Kentucky obstetrics clinics. This trial will provide evidence to evaluate this approach to delivering an established intervention in clinical practice.

The Investigators propose to test the effectiveness of the clinical intervention by using a two-armed cluster randomized controlled design. Eligible participants will be randomized to the intervention (ToPIC) or standard of care for smoking cessation in pregnancy. This pilot project will gather quantitative and qualitative data for a mixed-method, multi-stakeholder process evaluation of intervention training and delivery. Furthermore, the Investigators' use of Medicaid claims data to examine healthcare utilization outside of maternal and infant well-care visits will enhance understanding of the strengths and limitations of these data for future evaluations. This study has the potential to significantly impact the most vulnerable in Kentucky, where rates of tobacco use among pregnant women are among the highest in the nation.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* tobacco user
* able to read and write English
* Medicaid eligible

Exclusion Criteria:

* male

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — research participants must be pregnant
Enrollment: 66 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | Baseline to third trimester
  Change in urine cotinine level

SECONDARY OUTCOMES:
Number of cigarettes per day | Baseline to third trimester
  Self-reported change in number of cigarettes smoked per day
Smoking cessation after delivery | Prior to delivery hospitalization discharge, estimated 3 days
  Self-report smoking cessation
Infant birth weight | At time of delivery
  Infant weight measured in grams
Gestational age | At time of delivery
  Weeks of gestation at delivery
Health care utilization outside of well-visits | Birth to 6 months
  Maternal and infant visits for non-routine healthcare

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ashford, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky College of Nursing, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03442530/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03442530/Prot_SAP_001.pdf